CLINICAL TRIAL: NCT05821777
Title: A Phase 1/2a, First in Human, Open-Label, Multicenter, Dose Escalation Study With Expansion Cohorts to Evaluate the Safety, Tolerability, and Preliminary Activity of LB101 in Subjects With Advanced Solid Tumors
Brief Title: A Study to Evaluate Safety, Tolerability and Preliminary Activity of LB101 in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated the study due to non-safety reasons. Based on the data and the current competitive landscape, Sponsor made the decision to close the study.
Sponsor: Centessa Pharmaceuticals (UK) Limited (Industry)
Collaborators: LockBody Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Organization: Centessa Pharmaceuticals plc (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LB101-101; 2022-003928-40 (EudraCT Number)
Record Dates: First submitted 2023-03-17; First posted 2023-04-20 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: Part 1 of the study will be non-randomized and Part 2 design will depend on results of Part 1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LB101 (Experimental): Part 1
  Part 1a participants will receive LB101 once every 2 weeks (Q2W) (28-day cycle), with a preliminary plan for 6 sequential dose levels. Part 1b will be a dose optimization and will include >1 dose levels and/or dose schedules that have been deemed safe and tolerable in Part 1a.
  Part 2
  Dose regimen(s) for participants in Part 2 will be based on the results of Part 1.
  Interventions: Drug: LB101

INTERVENTIONS:
Drug: LB101 — Part 1: IV infusion of LB101 Q2W (28-day cycle) and Part 2: IV infusion of LB101

SUMMARY:
The purpose of this study is to assess safety, tolerability, and preliminary activity of LB101 monotherapy in participants with advanced solid tumors.

DETAILED DESCRIPTION:
This study consists of 2 parts: First in Human (FIH) dose escalation and dose optimization (Part 1a and Part 1b, respectively) and dose expansion (Part 2). Part 1 will evaluate LB101 monotherapy in participants with selected, advanced solid tumors and determine the Recommended Dose(s) for Expansion (RDE(s)) for Part 2. The design of Part 2 depends on the results of Part 1 and will further evaluate the safety, efficacy, tolerability, pharmacokinetics, and immune response of LB101.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants >= 18 years old
* Signed informed consent form (ICF)
* For Part 1: Participants who i). have a histologically confirmed solid tumor that is listed below and is advanced, unresectable, and/or metastatic and ii). have no standard therapy, are not candidates for available standard therapy, or have failed systemic therapy due to lack of response, progression, or intolerance:
* Non-small cell lung cancer (NSCLC), which is known to be PD L1 positive (combined positive score [CPS] ≥ 1 or tumor proportion score [TPS] ≥ 1%) after having received pembrolizumab or other analog immune checkpoint inhibitor at any stage of their prior therapy I. Subjects with PD-L1 positive NSCLC with known genomic alterations for which targeted therapy is approved are not required to have been treated with pembrolizumab, etc. but must have received such approved targeted therapy. Genomic alternations include, but are not limited to, epidermal growth factor receptor [EGFR] and anaplastic lymphoma kinase [ALK]
* Head and neck squamous cell carcinoma or cervical cancer, which is known to be PD-L1-positive, after having received immune checkpoint inhibitor at any stage of their prior therapy
* Cutaneous squamous cell cancer after having received immune checkpoint inhibitor at any stage of their prior therapy
* Colorectal cancer with low level microsatellite instability (MSI-low) and/or microsatellite stable(MSS)
* Ovarian cancer which is platinum resistant or platinum refractory, with platinum free interval of less than 6 months, and without rapidly progressing disease in the investigator's judgment
* Gastric cancer which is known to be PD-L1 positive after having received pembrolizumab or other analog immune checkpoint inhibitor at any stage of their prior therapy
* Participants have measurable disease according to RECIST v1.1
* Available archived tumor tissue sample (Part 1a)
* In Part 1a backfill cohort(s), Part 1b, and Part 2, subjects must agree to undergo baseline tumor biopsy
* Participants have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Participants have adequate hematological function
* Participants have adequate hepatic and renal function
* Participants have a baseline QT interval as corrected by Fridericia's formula <= 480 milliseconds
* Participants with life expectancy >= 12 weeks
* Participants have a body weight >= 40 kilograms
* For female participants of childbearing potential:
* Negative urine or serum pregnancy test
* Willing to use 2 highly effective methods of contraception
* For male participants who can father a child:
* Willing to use 2 highly effective methods of contraception

Exclusion Criteria:

* Participants with unknown PD-L1 status for the following tumor types: NSCLC, head and neck squamous cell carcinoma, or cervical cancer

  a.In Part 1a backfill cohort(s), any subject with unknown PD-L1 status
* Participants with known negative PD-L1 status
* Participants with NSCLC, head and neck squamous cell carcinoma, cervical cancer, cutaneous squamous cell cancer, or gastric cancer that have NOT received checkpoint inhibitor for advanced/metastatic disease, unless such therapy is not approved for treating a subject's specific condition
* Participants who receive adjuvant systemic therapy and progressed with advanced disease within 6 months of completing treatment
* Participants who have had previous exposure to CD47 or SIRPα targeting anticancer therapy
* Participants participating in another interventional clinical study
* Participants who have ongoing side effects to any prior therapy or procedure, which have not recovered to NCI CTCAE Grade <= 1
* Participants who have received immunosuppressive drugs within 7 days prior to the start of LB101 or systemic glucocorticoids equivalent
* Participants who have received a live attenuated vaccine within 4 weeks prior to the start of LB101. For any subject receiving an approved severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccine, the investigator will be advised to follow the vaccine label and/or local guidance
* Participants with primary brain tumors and evidence of new or progressing cerebrospinal or leptomeningeal metastases
* Participants who have a history of Grade ≥ 3 allergic reactions to monoclonal antibody therapy as well as known or suspected allergy or intolerance to any components of LB101
* Participants with active or suspected systemic inflammatory autoimmune diseases or with a history of documented autoimmune disease over the past 2 years
* Participants who have ongoing or active infection requiring IV anti-infective medications
* Participants with a known history of:
* Seropositivity for human immunodeficiency virus (HIV)
* Positive serology for hepatitis B, known history/positive serology for hepatitis C virus (HCV)
* Allogenic organ transplantation and/or hematopoietic stem cell transplantation
* Participants who have had a history of life-threatening treatment-related AEs with prior immunotherapy or who have not recovered from prior cancer therapy-induced AEs
* Participants with clinically significant ascites
* Participants with moderate bilateral pleural effusion or massive bilateral pleural effusion or respiratory dysfunction requiring drainage
* Participants with uncontrolled cardiovascular disease
* Participants with any other acute or chronic diseases, psychiatric disorders, or abnormal laboratory test values that, at the discretion of the investigators are deemed ineligible to participate
* Participants with a history of other advanced solid tumor malignancies except:
* Cured malignant tumors for > 2 years prior to enrollment and no known active disease
* Tumors with negligible risk of metastases or death
* Pregnant or lactating female participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Dose Limiting Toxicities (DLTs) as graded according to the NCI CTCAE v5.0 | 28 days following the first dose of LB101 (Days 1 to 28 of Cycle 1)
Part 1 and 2: Number of Participants with Treatment-Emergent Adverse Events (TEAEs) as defined as events that started or worsened after first dose of study intervention until 30 days after last dose | From start of study treatment up to 3 years
Part 1: Number of Participants with Recommended Dose(s) for Expansion | 28 days following the first dose of LB101 (Days 1 to 28 of Cycle 1)
  Recommended Dose for expansion will be determined.
Part 2: Proportion of Participants with Confirmed Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Evaluated by the Blinded Independent Central Review (BICR) | Up to 3 years

SECONDARY OUTCOMES:
Part 1 and 2: Proportion of Participants with Objective Response Rate (ORR) According to RECIST v1.1 Evaluated by the Investigator | Up to 3 years
Part 1 and 2: Duration of Response (DoR) According to RECIST v1.1 Evaluated by the Blinded Independent Central Review (BICR) | Time from first objective response to first occurrence of objective tumor progression or death from any cause (up to 3 years)
Part 1 and 2: Proportion of Participants with Disease Control Rate (DCR) According to RECIST v1.1 Evaluated by the Blinded Independent Central Review (BICR) | Up to 3 years
Part 1 and 2: Duration of Response (DoR) Assessed by Investigator | Time from first objective response to first occurrence of objective tumor progression or death from any cause (up to 3 years)
Part 1 and 2: Disease Control Rate (DCR) Assessed by Investigator | Up to 3 years
Part 1 and 2: Number of Participants with Antidrug Antibodies (ADA) and Neutralizing Antibodies (NAb) to LB101 | Up to 3 years
Part 1: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 2, 3, 5, 8, 11, 15, 16, and 22), Cycle 2 (Day 1, 2, 8, and 15), Cycle 3 (Day 1, and 15), and Cycle 4 (Day 1, and 15)
Part 2: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 15, 16, and 22), Cycle 2 (Day 1, and 15), and Cycle 3 (Day 1, and 15)
Part 1: Maximum (peak) Concentration (Cmax) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 2, 3, 5, 8, 11, 15, 16, and 22), Cycle 2 (Day 1, 2, 8, and 15), Cycle 3 (Day 1, and 15), and Cycle 4 (Day 1, and 15)
Part 2: Maximum (peak) Concentration (Cmax) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 15, 16, and 22), Cycle 2 (Day 1, and 15), and Cycle 3 (Day 1, and 15)
Part 1: Time to Maximum Observed Concentration (Tmax) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 2, 3, 5, 8, 11, 15, 16, and 22), Cycle 2 (Day 1, 2, 8, and 15), Cycle 3 (Day 1, and 15), and Cycle 4 (Day 1, and 15)
Part 2: Time to Maximum Observed Concentration (Tmax) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 15, 16, and 22), Cycle 2 (Day 1, and 15), and Cycle 3 (Day 1, and 15)
Part 1: Area Under the Concentration-time Curve at 14 days Post Drug Administration (AUC14days) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 2, 3, 5, 8, 11), Cycle 2 (Day 1, 2, and 8), Cycle 3 (Day 1), and Cycle 4 (Day 1)
Part 2: Area Under the Concentration-time Curve at 14 days Post Drug Administration (AUC14days) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1), Cycle 2 (Day 1), and Cycle 3 (Day 1)
Part 1: Area Under the Concentration-time Curve From Time 0 to the Last Quantifiable Concentration (AUC0-last) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 2, 3, 5, 8, 11, 15, 16, and 22), Cycle 2 (Day 1, 2, 8, and 15), Cycle 3 (Day 1, and 15), and Cycle 4 (Day 1, and 15)
Part 2: Area Under the Concentration-time Curve From Time 0 to the Last Quantifiable Concentration (AUC0-last) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 15, 16, and 22), Cycle 2 (Day 1, and 15), and Cycle 3 (Day 1, and 15)
Part 1: Elimination Half-life (t1/2) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 2, 3, 5, 8, 11, 15, 16, and 22), Cycle 2 (Day 1, 2, 8, and 15), Cycle 3 (Day 1, and 15), and Cycle 4 (Day 1, and 15)
Part 2: Elimination Half-life (t1/2) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 15, 16, and 22), Cycle 2 (Day 1, and 15), and Cycle 3 (Day 1, and 15)
Part 1: Elimination Rate Constant (Kel) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 2, 3, 5, 8, 11, 15, 16, and 22), Cycle 2 (Day 1, 2, 8, and 15), Cycle 3 (Day 1, and 15), and Cycle 4 (Day 1, and 15)
Part 2: Elimination Rate Constant (Kel) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 15, 16, and 22), Cycle 2 (Day 1, and 15), and Cycle 3 (Day 1, and 15)
Part 1: Apparent Total Body Clearance (CL/F) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 2, 3, 5, 8, 11, 15, 16, and 22), Cycle 2 (Day 1, 2, 8, and 15), Cycle 3 (Day 1, and 15), and Cycle 4 (Day 1, and 15)
Part 2: Apparent Total Body Clearance (CL/F) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 15, 16, and 22), Cycle 2 (Day 1, and 15), and Cycle 3 (Day 1, and 15)
Part 1: Apparent Volume of Distribution (Vd/F) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 2, 3, 5, 8, 11, 15, 16, and 22), Cycle 2 (Day 1, 2, 8, and 15), Cycle 3 (Day 1, and 15), and Cycle 4 (Day 1, and 15)
Part 2: Apparent Volume of Distribution (Vd/F) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 15, 16, and 22), Cycle 2 (Day 1, and 15), and Cycle 3 (Day 1, and 15)
Part 1: Predose Trough Concentrations (CTrough) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 2, 3, 5, 8, 11, 15, 16, and 22), Cycle 2 (Day 1, 2, 8, and 15), Cycle 3 (Day 1, and 15), and Cycle 4 (Day 1, and 15)
Part 2: Predose Trough Concentrations (CTrough) of LB101 | Day 0 (pre-dose) and at multiple time points (up to End of infusion) post-dose in Cycle 1 (Day 1, 15, 16, and 22), Cycle 2 (Day 1, and 15), and Cycle 3 (Day 1, and 15)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Sarah Cannon Research Institute at HealthONE., Denver, Colorado
  - Sarah Cannon Research Institute at Florida Cancer Specialists, Sarasota, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute at Tennessee Oncology Nashville, Nashville, Tennessee
  - NEXT Oncology - Dallas, Irving, Texas
  - NEXT Oncology, San Antonio, Texas
- Institut Gustave Roussy, Villejuif, France